CLINICAL TRIAL: NCT00457431
Title: Hypothermia After In-hospital Cardiac Arrest
Acronym: HACAinhospital
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: interim analysis with stopping for futility
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: University of Hamburg-Eppendorf (Other); University of Leipzig (Other); University of Jena (Other)
Responsible Party: Principal Investigator, Sebastian Wolfrum, D. Sebastian Wolfrum, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HACA in-hospital
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Cardiac Arrest
Keywords: in-hospital cardiac arrest; resuscitation; mild therapeutic hypothermia
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Standard therapy as used in the hospital's ICU
- Hypothermia (Active Comparator): Standard therapy as used in the hospital's ICU plus Hypothermia
  Interventions: Procedure: Mild therapeutic hypothermia

INTERVENTIONS:
Procedure: Mild therapeutic hypothermia — Mild therapeutic hypothermia will be performed by any methods applicable in the hospitals
  Arms: Hypothermia

SUMMARY:
ILCOR Recommendations "On the basis of the published evidence to date, the Advanced Life Support (ALS) Task Force of the International Liaison Committee on Resuscitation (ILCOR) made the following recommendations in October 2002: Unconscious adult patients with spontaneous circulation after out-of-hospital cardiac arrest should be cooled to 32°C to 34°C for 12 to 24 hours when the initial rhythm was ventricular fibrillation (VF).Such cooling may also be beneficial for other rhythms or in-hospital cardiac arrest" (Circulation. 2003;108:118-121). This study ist to investigate the efficacy of mild therapeutic hypothermia on mortality and neurological outcome in patients after in-hospital cardiac arrest.

DETAILED DESCRIPTION:
This is a randomized controlled multicenter trial. Patients after in-hospital cardiac arrest are randomized either to standard therapy or to standard therapy in addition to mild therapeutic hypothermia. Mild therapeutic hypothermia is performed for 24 hours with a target temperature of 32-34°C. Inclusion criteria are: Adult patients which have been resuscitated after cardiac arrest in-hospital and who remain unconscious after restoration of spontanous circulation. Exclusion criteria are: severe cardiogenic shock, severe rhythm disorders, major surgery within the last 10 days, planned surgery within the next 24 hours afer resuscitation, active bleeding, suspicion od intracranial bleeding, severe infection, such as pneumonia or sepsis, a severe neurological deficit before cardiac arrest, an aquired immun deficency, pregnacy. The primary endpoint is mortality for all causes after six months. Secondary endpoints are neurological outcome after six months measured by the Glasgow-Pittsburgh Cerebral Performance scale, and in-hospital-mortality.

ELIGIBILITY:
Inclusion Criteria:

* in-hospital cardiac arrest
* restoration of spontanous circulation
* unconsciousness
* age over 18
* initiation of mild therapeutic hypothermia is possible within 4h after resuscitation

Exclusion Criteria:

* active bleeding
* suspicion of intra cranial bleeding
* severe infection
* aquired immun deficency
* severe rhythm disorders
* suspicion of cerebral insult
* known severe cognotive deficit before the index event
* pregnancy
* pre existing disease which makes 6 months survival unlikely

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2007-04-03 (Actual); Primary Completion 2014-11-09 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
all cause mortality at 6 months | 6 months

SECONDARY OUTCOMES:
neurological outcome at six months measured by the Glasgow-Pittsburgh cerebral performance scale | 6 months
in-hospital all cause mortality | time until discharge or death

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Wolfrum, MD, Principal Investigator — University of Schleswig-Holstein, Campus Luebeck, Medical Clinic II
Locations (1):
- Sebastian Wolfrum, Lübeck, Schleswig-Holstein, Germany

REFERENCES:
- [Derived] Wolfrum S, Roedl K, Hanebutte A, Pfeifer R, Kurowski V, Riessen R, Daubmann A, Braune S, Soffker G, Bibiza-Freiwald E, Wegscheider K, Schunkert H, Thiele H, Kluge S; Hypothermia After In-Hospital Cardiac Arrest Study Group. Temperature Control After In-Hospital Cardiac Arrest: A Randomized Clinical Trial. Circulation. 2022 Nov;146(18):1357-1366. doi: 10.1161/CIRCULATIONAHA.122.060106. Epub 2022 Sep 28. PMID 36168956
- [Derived] Soar J, Nolan JP. Mild hypothermia for post cardiac arrest syndrome. BMJ. 2007 Sep 8;335(7618):459-60. doi: 10.1136/bmj.39315.519201.BE. PMID 17823147